CLINICAL TRIAL: NCT02515721
Title: Probe-based Confocal Laser Endomicroscopy for the Diagnosis of Gastric Intestinal Metaplasia,Intraepithelial Neoplasia,and Carcinoma:A Multicenter,Randomized,Controlled Trial
Brief Title: PCLE for the Diagnosis of Gastric Intestinal Metaplasia, Intraepithelial Neoplasia, and Carcinoma
Acronym: PCLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); Zhejiang University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Chief of the department of Gastroenterology, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2015SDU-QILU-G06
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Diagnostic Yield of Gastric Neoplasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pCLE-TB (Experimental): Patients will receive white-light endoscopic imaging, followed by probe-based Confocal Laser Endomicroscopy scanning on suspected lesions and 5 standardized locations. Then targeted Biopsies will be performed on locations with intestinal metaplasia, intraepithelial neoplasia, and carcinoma.
  Interventions: Device: pCLE-TB
- Virtual Chromoendoscopy -SB (Experimental): Patients will receive virtual chromoendoscopy using iScan. Standard biopsies will be performed on all suspected lesions and standardized loctaions.
  Interventions: Device: virtual chromoendoscopy-TB

INTERVENTIONS:
Device: pCLE-TB — Patients will receive white-light endoscopic imaging, followed by probe-based Confocal Laser Endomicroscopy scanning on suspected lesions and 5 standardized locations. Then targeted Biopsies will be performed on locations with intestinal metaplasia, intraepithelial neoplasia, and carcinoma.
  Other Names: probe-based confocal laser endomicroscopy with targeted biopsies
  Arms: pCLE-TB
Device: virtual chromoendoscopy-TB — Patients will receive virtual chromoendoscopy using iScan. Standard biopsies will be performed on all suspected lesions and standardized loctaions.
  Other Names: virtual chromoendoscopy with targeted biopsies
  Arms: Virtual Chromoendoscopy -SB

SUMMARY:
Early detection of gastric intestinal metaplasia (GIM) intraepithelial neoplasia (IN), and gastric cancer are essential to improve patients' outcomes. This study aims to compare the diagnostic yield of GIM, IN and early gastric cancer (EGC) by iScan combined probe-based confocal laser endomicroscopy (pCLE) and iScan alone.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80;
* patients with previous pathologic diagnosis of atrophic gastritis, gastric intestinal metaplasia, and low-grade intraepithelial neoplasia;
* agree to give written informed consent.

Exclusion Criteria:

* Patients with gastrectomy, acute GI bleeding, and known gastric neoplasia;
* Patients under conditions unsuitable for performing CLE including coagulopathy (prothrombin time <50% of control, partial thromboplastin time >50 s), impaired renal function (creatinine level >1.2 mg/dL), pregnancy or breastfeeding, and known allergy to fluorescein sodium;
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
the diagnostic yield of intestinal metaplasia, intraepithelial neoplasia, and gastric cancer | 12 months

SECONDARY OUTCOMES:
the biopsy number needed for diagnosis | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic unit of Qilu Hospital Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Zuo XL, Li Z, Li CQ, Zheng YY, Xu LD, Chen J, Lin R, Song J, Yu CH, Yue M, Zhou Q, Liu ZY, Li YQ. Probe-based endomicroscopy for in vivo detection of gastric intestinal metaplasia and neoplasia: a multicenter randomized controlled trial. Endoscopy. 2017 Nov;49(11):1033-1042. doi: 10.1055/s-0043-115382. Epub 2017 Jul 28. PMID 28753702